CLINICAL TRIAL: NCT04453644
Title: Effects of Stretching on Strength of Proximal and Distal Group of Muscles - A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RRC-2019-06
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: STRETCHING
Keywords: Muscle strength; muscle stretching exercises; strain gauge
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Hamstrings) (Experimental): Hamstring stretching would be done then isometric strength would be measured.
  Interventions: Other: Muscle static stretching
- Group B (Calf) (Experimental): Calf stretching would be done then isometric strength would be measured.
  Interventions: Other: Muscle static stretching

INTERVENTIONS:
Other: Muscle static stretching — On day-I: Static Stretching done for 2 minutes (SS2), on day-II: Static Stretching done for 4 minutes (SS4), and on day-III: Static Stretching done for 8 minutes (SS8).

SUMMARY:
Muscular flexibility is believed to prevent injuries and improve movement therefore most coaches include stretching exercises in their pre-competition and pre-exercise warm-up routines. One question arises here, should sports persons avoid stretching exercises prior to sporting events thereby exposing themselves to musculoskeletal injuries, or should they continue stretching exercises prior to sporting events and risk losing the maximal performance? The aim of this study is to compare the effects of 2, 4, and 8 min of static stretching (SS) on isometric maximum voluntary contraction (MVCF) force between proximal (Hamstrings) and distal group (Calf) of muscles.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the effects of 2, 4, and 8 min of static stretching (SS) on isometric maximum voluntary contraction (MVCF) force between proximal (Hamstrings) and distal group (Calf) of muscles.

DESIGN: Two-group pretest-posttest experimental design. METHODS: Each subject visited the Rehabilitation center on three days: On day-I for static stretching for 2 minutes (SS2), day-II for 4 minutes (SS4), and day-III for 8 minutes (SS8). Isometric Maximum Voluntary Contraction Force (MVCF) measurement was done prior (Pre), 0-min, 10-min, and 20-min post-intervention (i.e. stretching). Each visit was separated by a gap of at least 3-4 days. On each visit, each subject underwent (a). Pre-intervention evaluation, (b). Intervention, (c). Post-intervention evaluation. Subjects performed stretching exercises under the supervision of expert Physical Therapist. The outcome assessor who was kept blind to study protocol did all measurements.

ELIGIBILITY:
Inclusion Criteria:

For group A: subjects performed active knee extension test and those lacking at least 20 degrees of active knee extension range, with hip in 90 degree of flexion were selected. For group B (Calf): Subjects performed active foot dorsiflexion in long sitting position with back supported against the wall and those having not more than 20-degree range of motion were selected.

Selected subjects used to engage in 1-5 hours of regular physical activity per week (recreationally active) that does not involve stretching exercise

Exclusion Criteria:

Subjects reporting any current or ongoing neuromuscular disease, injury specific to lower limb joints, any apparent limit in knee or ankle ROM and competitive/professional athletes were excluded from study.

Ages: 22 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Change in isometric maximum voluntary contraction force before and after stretching | MVCF was measured immediately (0 min), 10-min and 20 min post intervention on 3 different days, with each day separated by gap of 3-4 days.
  Change in isometric muscle strength measured before and after stretching using strain gauge on 3 different days

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alghadir AH, Khan M, Quddus N, Chawla C. Effects of different stretch durations on the strength of the proximal and distal group of muscles - a randomized trial. Medicine (Baltimore). 2022 Oct 28;101(43):e31279. doi: 10.1097/MD.0000000000031279. PMID 36316911